CLINICAL TRIAL: NCT03643159
Title: A Multicenter, 180-day Pragmatic Clinical Trial to Measure the Difference in All-cause Hospitalizations for Patients Who Are Using Abilify MyCite Versus Virtual Matched Controls in Adults With Schizophrenia, Bipolar 1 Disorder, and Major Depressive Disorder
Brief Title: A Trial to Measure the Difference in All-cause Hospitalizations for Participants Who Are Using Abilify MyCite Versus Virtual Matched Controls in Adults With Schizophrenia, Bipolar 1 Disorder, and Major Depressive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in participant recruitment
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 316-13-217
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Bipolar 1 Disorder; Major Depressive Disorder
Keywords: Digital Medicine System
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Abilify MyCite (Experimental): Participants received Abilify MyCite during Months 1-3. During Months 4-6 use of Abilify MyCite was to be prohibited. Thereafter, at Day 180, a second, optional interventional period (up to 6 months of Abilify MyCite) could have been initiated per the joint decision of the participants with their study physician.
  Interventions: Combination Product: Abilify MyCite - Digital Medicine System; Drug: Aripiprazole or other oral antipsychotics
- Virtual Matched Controls (Active Comparator): Virtual matched controls were to receive treatment as usual (that is, any product other than Abilify MyCite, which could have been oral aripiprazole or any other product) throughout the duration of the trial. Virtual matched controls were not to be enrolled into the study, but identified from health insurance claims data and matched to the enrolled Abilify MyCite participants at the end of the study for analysis.
  Interventions: Drug: Aripiprazole or other oral antipsychotics

INTERVENTIONS:
Combination Product: Abilify MyCite - Digital Medicine System — The Abilify MyCite system is a drug-device combination product comprised of aripiprazole (an atypical antipsychotic) tablets embedded with a sensor that communicates with a patch (wearable sensor) and a medical software application with collected information (ingestion, mood, activity, rest) tracked and summarized for participants, healthcare providers, and potential caregivers. Abilify MyCite is intended to track drug ingestion and is indicated for the treatment of adults with schizophrenia (SCH), bipolar 1 disorder (BP1) (acute treatment of adults with manic and mixed episodes or maintenance treatment of adults), and adjunctive treatment of adults with major depressive disorder (MDD).
  Arms: Abilify MyCite
Drug: Aripiprazole or other oral antipsychotics — For the treatment of adults with SCH, BP1 (acute treatment of adults with manic and mixed episodes or maintenance treatment of adults), and adjunctive treatment of adults with MDD.

SUMMARY:
The primary objective of this pragmatic clinical trial (Main Study) was to assess the difference between all-cause hospitalizations in participants using Abilify MyCite versus virtual matched controls. In addition, secondary and exploratory objectives were to assess medication adherence, healthcare utilization and costs, and patient-reported outcomes.

DETAILED DESCRIPTION:
This was a phase 4, open-label, prospective, pragmatic clinical trial to assess the difference between all-cause hospitalizations in participants using Abilify MyCite (for Months 1-3, then prohibited for Months 4-6) versus virtual matched controls from baseline to Day 180. Virtual matched controls were to receive treatment as usual (that is, any product other than Abilify MyCite, which was oral aripiprazole or any other product). Eligible participants entered a screening period of up to 13 days. For participants enrolling into the study, those not on aripiprazole at screening used the screening period for conversion to aripiprazole from other antipsychotics. Virtual matched controls were not to be enrolled into the study, but identified from health insurance claims data and matched to the enrolled Abilify MyCite participants at the end of the study for analysis.

After the visit at Day 180, a second, optional interventional period (up to 6 months of Abilify MyCite) could have been initiated per the joint decision of the participants with their study physician; participants in this second, optional interventional period were to have a visit at Day 360. During this second, optional interventional period, participants may have started and stopped Abilify MyCite as clinically indicated.

A parallel exploratory study that would utilize a different set of physicians and participants from the main study was planned; however, that study was never initiated.

ELIGIBILITY:
Inclusion Criteria:

* Participants are actively enrolled in an Anthem-affiliated commercial, Medicaid, or Medicare health plan with medical and pharmacy benefits.
* Participants must have a smartphone with data plan.
* Participants currently prescribed aripiprazole, or appropriate for aripiprazole treatment.
* Participants must have a current diagnosis of SCH, BP1, or MDD.

Exclusion Criteria:

* Any participant who participated in another clinical trial within 30 days of enrollment into the current study.
* Females who are breast-feeding and/or who are pregnant at the time of study enrollment, or who plan to become pregnant during the study.
* Participants who are currently being treated with a long-acting injectable antipsychotic.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Siyan Clinical Research, Santa Rosa, California
  - Psychiatric Addiction Curative/PACT Atlanta LLC, Decatur, Georgia
  - Georgia Psychiatry and Sleep, Smyrna, Georgia
  - Kolade Research Institute, Las Vegas, Nevada
  - Signature Research Associates, Inc., Fairlawn, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Virtual matched controls were not to be enrolled into the study, but identified from health insurance claims data and matched to the enrolled Abilify MyCite participants at the end of the study for analysis. Since the study was terminated early, no matching occurred.
Groups:
- Abilify MyCite: Participants received Abilify MyCite during Months 1-3. The treatment medication dose decision was determined by the study physicians independent from the protocol.
Period: Overall Study
Arm/Group | Abilify MyCite
Started | 2
Received At Least 1 Dose Of Study Drug | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety: All participants who received at least 1 dose of Abilify MyCite or who were a virtual matched control.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abilify MyCite | Virtual Matched Controls | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.

OUTCOME MEASURES:

1. Primary Outcome: Difference In The Number Of Participants With All-cause Hospitalizations For Participants Using Abilify MyCite Versus Virtual Matched Controls From Baseline To Day 180
Description: This outcome measure describes the difference in all-cause hospitalizations (that is hospitalizations for any reason) between the number of participants using Abilify MyCite and those receiving treatment as usual (the virtual matched controls). Due to early study termination, efficacy data were not collected.
Time Frame: Baseline through Day 180
Population: Efficacy Analysis: All participants who received at least 1 dose of Abilify MyCite or who were a virtual matched control and had efficacy data. Both participants were excluded from efficacy analysis because they discontinued study therapy early. In addition, efficacy data were not collected due to early study termination.
Arm/Group | Abilify MyCite | Virtual Matched Controls
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Difference In The Number Of Participants With At Least 80% Proportion Of Days Covered (PDC) (With Antipsychotic Medication) For Participants Using Abilify MyCite Versus Virtual Matched Controls From Baseline To Day 180
Description: This outcome measure describes the difference in the number of participants with at least 80% PDC (with antipsychotic medication) between those using Abilify MyCite and those receiving treatment as usual (the virtual matched controls). Due to early study termination, efficacy data were not collected.
Time Frame: Baseline through Day 180
Population: as for outcome 1
Arm/Group | Abilify MyCite | Virtual Matched Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) to Day 49
Description: The 2 enrolled participants both received Abilify MyCite. According to protocol, serious and other adverse events were not to be assessed for Virtual Matched Controls.
Arm/Group | Abilify MyCite
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abilify MyCite (N=2)
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor due to difficulty in participant recruitment, leading to a small number of participants enrolled. Due to early termination of the study, no efficacy data were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review, edit, and authorize publications.

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03643159/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03643159/SAP_001.pdf